CLINICAL TRIAL: NCT02065700
Title: A Multicenter, Open-label, Long-term Follow-up Safety and Efficacy Study of GLPG0634 Treatment in Subjects With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: Long-term Follow-up Study of GLPG0634 in Active Rheumatoid Arthritis Participants
Acronym: DARWIN3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-205; 2012-003655-11 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; insufficient responders
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Filgotinib Darwin 1 (Experimental): Participants in Study GLPG0634-CL-203 (NCT01888874) were rolled-over to receive an oral dose of filgotinib at a daily dose of 200 milligrams (mg) in this extension study, with the exception of male participants in the United States (US) who were limited to a daily dose of 100 mg due to a Food and Drug Administration (FDA) requirement based on a non-clinical finding. Treatment was administered until marketing, local (if applicable) regulatory and/or pertinent local reimbursement approval.
  In case of intolerance or for safety reasons, and as per investigator's discretion, a daily dose of filgotinib 200 mg could be decreased to 100 mg per day, and later returned to 200 mg per day after the reasons for decreasing the dose were resolved.
  Interventions: Drug: Filgotinib
- Filgotinib Darwin 2 (Experimental): Participants from Study GLPG0634-CL-204 (NCT01894516) were rolled-over to receive oral dose of filgotinib tablet at 200 mg once daily (q.d) in this extension study. Treatment was administered until marketing, local (if applicable) regulatory and/or pertinent local reimbursement approval.
  Participants started the study with the same dose level (filgotinib 200 mg per day) and in case of intolerance or safety reasons and as per investigator's discretion, the daily dose of filgotinib was decreased to 100 mg q.d and was returned to 200 mg per day after the reasons for decreasing the dose had resolved and at the investigator's discretion.
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Administered as Oral Tablets
  Other Names: GS-6034; GLPG0634

SUMMARY:
The primary objective of the study was to evaluate the long-term safety and tolerability of filgotinib (formerly GLPG0634) for the treatment of rheumatoid arthritis.

Participants were enrolled in this open-label long-term follow-up study after they had completed one of the two core studies, GLPG0634-CL-203 (DARWIN1) (NCT01888874) or GLPG0634-CL-204 (DARWIN2) (NCT01894516), and were evaluated for any side effects that might have occured (long-term safety and tolerability) when taking filgotinib. During the course of the study, participants were also examined for long-term effects of filgotinib administration on disease activity (efficacy), participant's disability, fatigue, and quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who completed one of the qualifying core studies GLPG0634-CL-203 or GLPG0634-CL-204 and may benefit from filgotinib long-term treatment according to the Investigator's judgment
* Females of childbearing potential and sexually active men must agree to use highly effective method of birth control as specified in the protocol, during the study and for at least 12 weeks after the last dose of filgotinib

Key Exclusion Criteria:

* Participants who prematurely withdrew from one of the 2 core studies (GLPG0634-CL-203 or GLPG0634-CL-204), for any reason
* Persistent abnormal lab values during one of the 2 core studies (GLPG0634-CL-203 or GLPG0634-CL-204), according to the Investigator's judgment
* Diagnosis of rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis, except for secondary Sjogren's syndrome
* Any condition or circumstances which, in the opinion of the Investigator, may make a participant unlikely or unable to complete the study or comply with study procedures and requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (111):
- United States (15):
  - Arthro, Arthritis Care & Research, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Mesa, Arizona
  - C.V. Mehta MD Medical Corp., Hemet, California
  - Desert Medical Advances, Palm Desert, California
  - RASF Clinical Research Center, Boca Raton, Florida
  - Millenium Research, Ormond Beach, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Springfield Clinic, Springfield, Illinois
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Physicians East, Greenville, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Low County Rheumatology PA, Charleston, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Austin Rheumatology Research PA, Austin, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
- Argentina (8):
  - Atencion Integral en Reumatologa, Buenos Aires
  - CER Intituto Medico, Buenos Aires
  - Organizacion Medica de Investigaciones (OMI), Buenos Aires
  - Instituto Reumatologico Strusberg, Córdoba
  - CIMeL Centro dee Investigacion Medico Lanus, Lanús
  - Instituto CAICI, Rosario
  - Instituto de Asistencia Reumatologia Integral - IARI, San Fernando
  - Centro Médico Privado de Reumatologia, San Miguel de Tucumán
- Australia (3):
  - Flinders Medical Centre, Bedford Park, Flinders Drive, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven, Leuven
- Bulgaria (5):
  - University "Multiprofile Hospital for Active Treatment - Kaspela" LTD, Plovdiv
  - Multiprofile Hospital for Active Treatment - Ruse, Rousse
  - Diagnostic Consultative Center "Sveta Anna" LTD, Sofia
  - National Multiprofile Transport Hospital "Tsar Boris III," Sofia, Clinical of Internal Diseases, Sofia
  - University Multiprofile Hospital for Active Treatment "SV. Ivan Rilski" EAD, Sofia, Rheumatology Clinic, Sofia
- Chile (5):
  - Hospital Regional "Guillermo Grant Benavente", Santiago
  - Prosalud, Santiago
  - Someal SA, Santiago
  - Centro de Investigacion Clinica del Sur, Temuco
  - Consulta Privada Dra. Ponce, Temuco
- Colombia (7):
  - Medicity S.A.S., Bucaramanga, Santander Department
  - Circaribe S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas (CIREEM), Bogotá
  - Riesgo De Fractura Cayre Ips7, Bogotá
  - Idearg Sas, Bogotá
  - Preventive Care SAS, Cundinamarca
  - Hospital Pablo Tobon Uribe, Medellín
- Czechia (4):
  - Revmatologie S.R.O, Brno
  - Revmatologicka a interni ambulance, Kladno
  - Revmatologicka ambulance, Praha-Nusle
  - PV-Medical S.R.O., Zlín
- Hospitaux de Hautepierre, Strasbourg, France
- Germany (2):
  - Schlossparkklinik - Akad. Lehrkrankenhaus Charite, Berlin
  - MVZ Rheumatologie and Autoimmun Medizin HH GmbH, Hamburg
- Guatemala (6):
  - Centro Clinico, Guatemala City
  - Clinica de Especialidades Medicas, Guatemala City
  - Clinica Medica Especializada en Reumatologia, Guatemala City
  - Clinica Medica, Guatemala City
  - Reuma S.A., Guatemala City
  - Reuma-Centro, Guatemala City
- Hungary (5):
  - Gyogyszervizs galo Kozpont Kft, Balatonfüred
  - QualiClinic Kft., Budapest
  - Reumatologiai Kft., Budapest
  - Markhot Ferenc Hospital, Rheumatology, Eger
  - Csolnoky Ferenc Hospital, Rheumatology, Veszprém
- Israel (2):
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
- Latvia (5):
  - Ltd M&M Centr, Ādaži
  - SIA Arijas Ancane's Family Doctor, Baldone
  - Daugavpils Regional Hospital, Daugavpils
  - L. Atikes doktorats, Liepāja
  - 'Bruninieku' polyclinic, Riga
- Mexico (7):
  - Centro de Estudios de Investigacion Basica y Clinica, SC, Guadalajara
  - Centro Medico Dalinde, Mexico City
  - Arke Estudios Clinicos S.A. de C.V., México
  - Clinstile, S.A. de C.V., México
  - Hospital General de México, México
  - Hospital Universitario José E. Gonzalez, Monterrey
  - OSMO, Oaxaca City
- IMSP Institutul de Cardiologie, Chisinau, Moldova
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Timaru Rheumatology Studies, Timaru
- Poland (11):
  - NZOZ Osteo-Medic s.c., Bialystok
  - Centrum Medyczne Silesiana Sp. Z.o.o., Bytom
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne Plejady, Krakow
  - NZOZ "DOBRY LEKARZ" Specjalistyczne Poradnie Lekarskie, Krakow
  - Specjalistyczne Centrum Medyczne Nowomed, Krakow
  - NZOZ Przychodnia Lekarska "Eskulap", Skierniewice
  - Powiatowy Zaklad Opieki Zdrowotnej w Starachowicach, Starachowice
  - NZOZ "Nasz Lekarz" Pratyka Grupowa Lekarzy Rodzinnychz, Torun
  - AMED Medical Center, Warsaw
  - Rheumatica Sp. Z.o.o., Warsaw
- Romania (2):
  - Spitalul Clinic Sfanta Maria, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Galati, Galati
- Russia (8):
  - First Moscow State Medical University n.a. I.M. Sechenova of the Ministry of Health, Moscow
  - Scientific Research Institute of Rheumatology, Moscow
  - City Clinical Hospital #5, Nizhny Novgorod
  - GBOU VPO Orenburg State Medical University, Orenburg
  - Ryazan State Medical University, Ryazan
  - City Hospital #26, Saint Petersburg
  - Regional Clinical Hospital, Saratov
  - Vladimir Regional State Instituion of Healthcare, Vladimir
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Sanatorio Nuestra Señora de la Esperanza, A Coruña
  - Hospital Parc Tauli, Sabadell
- Ukraine (7):
  - Communal Institution of Healthcare - Kharkiv City Clinical Hospital #13, Kharkiv
  - Kharkiv Medical Academy of Postgraduate Education, Department of Cardiology, Kharkiv
  - L.T. Malaya Therapy Institute of National Academy of Medical Sciences of Ukraine, Kharkiv
  - Kherson City Clinical Hospital N. A. Afanasii and Olga Tropin, Kherson
  - Municipal Non-Profit Institution Consultative and Diagnostic Centre of Desnyasky District of Kyiv, Kiev
  - Municipal Non-profit Enterprise Consultative and Diagnostic Center of Pechersk District of Kiev city, Kyiv
  - Vinnitsya Regional Clinical Hospital Named after M.I.Pirogov, Rheumatology Department, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for clinical trials that support an approved indication in the EU and the US for which Galapagos is the Marketing Authorisation / New Drug Application Holder, with a marketing authorisation date on or after January 1, 2021 and for which the summary results have been published on ClinicalTrials.gov (CT.gov) and/or the EU Clinical Trials Register (EU CTR). For clinical trials of newly approved compounds or indications the IPD can be requested at earliest 6 months after the EMA and FDA approval. The study last patient last visit (LPLV) must have occurred at least 18 months prior to the request.

REFERENCES:
- [Result] Genovese MC, Kavanaugh A, Winthrop K, et al. Long Term Safety of Filgotinib in the Treatment of Rheumatoid Arthritis: Week 84 Data from a Phase 2b Open-Label Extension Study [abstract]. Arthritis Rheumatol. 2017; 69 (suppl 10).
- [Result] Kavanaugh A, Westhovens R, Winthrop K, et al. Rheumatoid Arthritis Treatment with Filgotinib: Week 156 Safety and Efficacy Data from a Phase 2b Open-Label Extension Study [abstract]. Arthritis Rheumatol. 2019; 71 (suppl 10).
- [Result] R. Westhovens, R. Alten, K. Winthrop, et al. Long term safety of filgotinib in the treatment of rheumatoid arthritis: week 108 data from a phase 2b open-label extension study. [abstract]. Ann Rheum Dis. 2018;77 (suppl 2)
- [Result] Kavanaugh A, Genovese MC, Winthrop K, et al. Rheumatoid Arthritis Treatment with Filgotinib: Week 132 Safety Data from a Phase 2b Open-Label Extension Study [abstract]. Arthritis Rheumatol. 2018; 70 (suppl 9).
- [Result] Kavanaugh A, Westhovens RR, Winthrop KL, Lee SJ, Tan Y, An D, Ye L, Sundy JS, Besuyen R, Meuleners L, Stanislavchuk M, Spindler AJ, Greenwald M, Alten R, Genovese MC. Safety and Efficacy of Filgotinib: Up to 4-year Results From an Open-label Extension Study of Phase II Rheumatoid Arthritis Programs. J Rheumatol. 2021 Aug;48(8):1230-1238. doi: 10.3899/jrheum.201183. Epub 2021 Feb 1. PMID 33526618
- [Derived] Westhovens R, Winthrop KL, Kavanaugh A, Greenwald M, Dagna L, Cseuz R, Besuyen R, de Vries D, Modgill V, Le LH, Genovese MC, Emery P, Verschueren P, Alten R. Safety and efficacy of filgotinib in patients with rheumatoid arthritis: final results of the DARWIN 3 long-term extension study. RMD Open. 2025 Jan 30;11(1):e004857. doi: 10.1136/rmdopen-2024-004857. PMID 39884731
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active rheumatoid arthritis were enrolled in this study.
Pre-assignment Details: Participants from DARWIN1 or DARWIN2 were rolled over into this extension study. As per planned analysis, data was collected and analyzed based on the parent study i.e. DARWIN 1 and DARWIN 2. No comparison/collection/analysis was planned based on extension study dose as it was not considered meaningful.
Period: Overall Study
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Started | 497 | 242
Male US Participants | 7 | 0
Completed | 161 | 81
Not Completed | 336 | 161
Not completed — Adverse Event | 165 | 101
Not completed — Withdrawal by Subject | 90 | 29
Not completed — Lost to Follow-up | 12 | 9
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor Request | 38 | 15
Not completed — Treatment Failure | 3 | 2
Not completed — Use of Non-permitted Concurrent Therapy | 3 | 0
Not completed — Adverse Event and Treatment Failure | 0 | 2
Not completed — Non-compliance with Study Procedures | 2 | 0
Not completed — Not Defined | 21 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who enrolled in the extension study and received at least one dose of study drug. As prespecified in the protocol, data was collected and analyzed based on their originating parent study I.e. DARWIN 1 and DARWIN 2.
Groups:
- Filgotinib Darwin 1: Participants in Study GLPG0634-CL-203 (NCT01888874) were rolled-over to receive an oral dose of filgotinib at a daily dose of 200 mg in this extension study, with the exception of male participants in the US who were limited to a daily dose of 100 mg due to an FDA requirement based on a non-clinical finding. Treatment was administered until marketing, local (if applicable) regulatory and/or pertinent local reimbursement approval.
  In case of intolerance or for safety reasons, and as per investigator's discretion, a daily dose of filgotinib 200 mg could be decreased to 100 mg per day, and later returned to 200 mg per day after the reasons for decreasing the dose were resolved.
- Filgotinib Darwin 2: Participants from Study GLPG0634-CL-204 (NCT01894516) were rolled-over to receive oral dose of filgotinib tablet at 200 mg q.d in this extension study. Treatment was administered until marketing, local (if applicable) regulatory and/or pertinent local reimbursement approval.
  Participants started the study with the same dose level (filgotinib 200 mg per day) and in case of intolerance or safety reasons and as per investigator's discretion, the daily dose of filgotinib was decreased to 100 mg q.d and was returned to 200 mg per day after the reasons for decreasing the dose had resolved and at the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2 | Total
Number analyzed (Participants) | 497 | 242 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.7) | 52 (12.2) | 53 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 198 | 603
  Male | 92 | 44 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 208 | 85 | 293
  Not Hispanic or Latino | 289 | 157 | 446
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 374 | 181 | 555
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 119 | 56 | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events
Description: An Adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
  Treatment-emergent adverse events (TEAEs) were defined as any AEs with an onset date on or after the filgotinib start date in the core studies or GLPG0634-CL-205 (NCT02065700), and no later than 30 days after permanent discontinuation of filgotinib in GLPG0634-CL-205 (NCT02065700) or of either 30 days after the last dose date.
Time Frame: From First dose to Week 437
Population: Safety Analysis Set. As prespecified in the protocol, data was collected and analyzed based on their originating parent study i.e. DARWIN 1 and DARWIN 2.
Measure: Number; unit: participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
participants | 453 | 223

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Response: Non-Responder Imputation (NRI)
Description: The American College of Rheumatology (ACR) response was a measurement of improvement in multiple disease assessment criteria.
  The ACR20 response was defined as: 1) ≥ 20% improvement from baseline in swollen joint count 66 (SJC66), and 2) ≥ 20% improvement from baseline in tender joint count 68 (TJC68), and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain visual analog scale (VAS) (taken from the Health Assessment Questionnaire - Disability Index [HAQ-DI]), 2.Subject's Global Assessment of Disease Activity (SGA) (VAS), 3. Physician's Global Assessment of Disease Activity (PGA) (VAS), 4. Total HAQ-DI score, and 5. High-Sensitivity C- Reactive Protein (hsCRP).
Time Frame: Extension Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, 384, 396, 408
Population: The Full Analysis Set (FAS) included all participants who enrolled in the extension study and received at least one dose of study drug.
  NRI: Participants with missing outcomes were set as nonresponders for binary response measurements. As prespecified in the protocol, data was collected and analyzed based on their originating parent study i.e. DARWIN 1 and DARWIN 2.
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline | 76.5 | 77.3
  Week 12 | 83.9 | 83.1
  Week 24 | 75.3 | 77.7
  Week 36 | 75.1 | 75.2
  Week 48 | 71.8 | 71.1
  Week 60 | 67.8 | 69.4
  Week 72 | 68.4 | 62.4
  Week 84 | 65.8 | 64.5
  Week 96 | 68.2 | 61.6
  Week 108 | 61.6 | 58.3
  Week 120 | 57.7 | 59.1
  Week 132 | 59.0 | 57.4
  Week 144 | 56.3 | 57.4
  Week 156 | 50.7 | 50.4
  Week 168 | 52.3 | 47.9
  Week 180 | 52.1 | 51.7
  Week 192 | 49.7 | 48.8
  Week 204 | 48.9 | 50.8
  Week 216 | 45.7 | 50.8
  Week 228 | 47.9 | 48.3
  Week 240 | 45.5 | 43.8
  Week 252 | 42.1 | 42.1
  Week 264 | 39.4 | 40.9
  Week 276 | 39.6 | 44.2
  Week 288 | 36.6 | 38.8
  Week 300 | 35.6 | 39.7
  Week 312 | 36.8 | 36.0
  Week 324 | 36.6 | 37.2
  Week 336 | 34.6 | 35.5
  Week 348 | 33.2 | 34.7
  Week 360 | 31.4 | 31.4
  Week 372 | 30.0 | 28.9
  Week 384 | 28.0 | 27.7
  Week 396 | 26.2 | 28.5
  Week 408 | 0.4 | 0.4

3. Secondary Outcome: Percentage of Participants Achieving ACR20 Response: Observed Case (OC)
Description: The ACR response was a measurement of improvement in multiple disease assessment criteria.
  The ACR20 response was defined as: 1) ≥ 20% improvement from baseline in SJC66, and 2) ≥ 20% improvement from baseline in tender TJC68, and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2.SGA (VAS), 3. PGA (VAS), 4. Total HAQ-DI score, and 5. hsCRP.
Time Frame: as for outcome 2
Population: FAS with available data was analyzed. OC: only observed values were used for analysis. No missing data imputation was performed. Different participants could be analyzed at different timepoints, resulting in overall FAS participants being analyzed. As prespecified in the protocol, data was collected and analyzed based on their originating parent study i.e. DARWIN 1 and DARWIN 2.
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline: number analyzed (Participants) | 491 | 235
  Extension Baseline | 77.4 | 79.6
  Week 12: number analyzed (Participants) | 484 | 230
  Week 12 | 86.2 | 87.4
  Week 24: number analyzed (Participants) | 441 | 210
  Week 24 | 84.8 | 89.5
  Week 36: number analyzed (Participants) | 431 | 204
  Week 36 | 86.5 | 89.2
  Week 48: number analyzed (Participants) | 422 | 198
  Week 48 | 84.6 | 86.9
  Week 60: number analyzed (Participants) | 399 | 185
  Week 60 | 84.5 | 90.8
  Week 72: number analyzed (Participants) | 387 | 172
  Week 72 | 87.9 | 87.8
  Week 84: number analyzed (Participants) | 375 | 170
  Week 84 | 87.2 | 91.8
  Week 96: number analyzed (Participants) | 377 | 163
  Week 96 | 89.9 | 91.4
  Week 108: number analyzed (Participants) | 356 | 158
  Week 108 | 86.0 | 89.2
  Week 120: number analyzed (Participants) | 334 | 157
  Week 120 | 85.9 | 91.1
  Week 132: number analyzed (Participants) | 333 | 151
  Week 132 | 88.0 | 92.1
  Week 144: number analyzed (Participants) | 323 | 155
  Week 144 | 86.7 | 89.7
  Week 156: number analyzed (Participants) | 289 | 136
  Week 156 | 87.2 | 89.7
  Week 168: number analyzed (Participants) | 298 | 138
  Week 168 | 87.2 | 84.1
  Week 180: number analyzed (Participants) | 291 | 141
  Week 180 | 89.0 | 88.7
  Week 192: number analyzed (Participants) | 281 | 133
  Week 192 | 87.9 | 88.7
  Week 204: number analyzed (Participants) | 272 | 134
  Week 204 | 89.3 | 91.8
  Week 216: number analyzed (Participants) | 262 | 132
  Week 216 | 86.6 | 93.2
  Week 228: number analyzed (Participants) | 266 | 126
  Week 228 | 89.5 | 92.9
  Week 240: number analyzed (Participants) | 256 | 119
  Week 240 | 88.3 | 89.1
  Week 252: number analyzed (Participants) | 233 | 111
  Week 252 | 89.7 | 91.9
  Week 264: number analyzed (Participants) | 227 | 109
  Week 264 | 86.3 | 90.8
  Week 276: number analyzed (Participants) | 215 | 114
  Week 276 | 91.6 | 93.9
  Week 288: number analyzed (Participants) | 207 | 110
  Week 288 | 87.9 | 85.5
  Week 300: number analyzed (Participants) | 201 | 105
  Week 300 | 88.1 | 91.4
  Week 312: number analyzed (Participants) | 206 | 100
  Week 312 | 88.8 | 87.0
  Week 324: number analyzed (Participants) | 203 | 104
  Week 324 | 89.7 | 86.5
  Week 336: number analyzed (Participants) | 194 | 97
  Week 336 | 88.7 | 88.7
  Week 348: number analyzed (Participants) | 188 | 92
  Week 348 | 87.8 | 91.3
  Week 360: number analyzed (Participants) | 180 | 86
  Week 360 | 86.7 | 88.4
  Week 372: number analyzed (Participants) | 166 | 82
  Week 372 | 89.8 | 85.4
  Week 384: number analyzed (Participants) | 163 | 79
  Week 384 | 85.3 | 84.8
  Week 396: number analyzed (Participants) | 153 | 75
  Week 396 | 85.0 | 92.0
  Week 408: number analyzed (Participants) | 3 | 2
  Week 408 | 66.7 | 50.0

4. Secondary Outcome: Percentage of Participants Achieving ACR50 Response: NRI
Description: The ACR response was a measurement of improvement in multiple disease assessment criteria.
  ACR50 response was defined as: 1) ≥ 50% improvement from baseline in SJC66, and 2) ≥ 50% improvement from baseline in TJC68, and 3) ≥ 50% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI) 2.SGA (VAS) 3. PGA (VAS) 4. Total HAQ-DI score 5. hsCRP.
Time Frame: as for outcome 2
Population: FAS. NRI: Participants with missing outcomes were set as nonresponders for binary response measurements. As prespecified in the protocol, data was collected and analyzed based on their originating parent study i.e. DARWIN 1 and DARWIN 2.
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline | 48.5 | 45.0
  Week 12 | 60.8 | 61.2
  Week 24 | 56.7 | 60.3
  Week 36 | 58.1 | 60.3
  Week 48 | 55.9 | 53.7
  Week 60 | 53.9 | 51.2
  Week 72 | 53.3 | 47.1
  Week 84 | 52.9 | 51.7
  Week 96 | 55.5 | 47.1
  Week 108 | 49.1 | 43.8
  Week 120 | 48.7 | 43.8
  Week 132 | 47.5 | 42.1
  Week 144 | 46.9 | 43.0
  Week 156 | 42.3 | 35.1
  Week 168 | 43.9 | 34.7
  Week 180 | 42.7 | 38.8
  Week 192 | 38.4 | 37.6
  Week 204 | 37.8 | 38.4
  Week 216 | 36.0 | 35.1
  Week 228 | 38.4 | 34.7
  Week 240 | 34.2 | 33.9
  Week 252 | 32.0 | 32.6
  Week 264 | 30.6 | 33.1
  Week 276 | 29.6 | 36.0
  Week 288 | 29.8 | 33.5
  Week 300 | 29.2 | 28.9
  Week 312 | 29.0 | 26.9
  Week 324 | 30.0 | 28.1
  Week 336 | 27.4 | 25.6
  Week 348 | 27.2 | 26.4
  Week 360 | 24.5 | 24.0
  Week 372 | 23.7 | 24.4
  Week 384 | 21.3 | 21.5
  Week 396 | 19.9 | 20.7
  Week 408 | 0.4 | 0.4

5. Secondary Outcome: Percentage of Participants Achieving ACR50 Response: OC
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline: number analyzed (Participants) | 488 | 235
  Extension Baseline | 49.4 | 46.4
  Week 12: number analyzed (Participants) | 484 | 231
  Week 12 | 62.4 | 64.1
  Week 24: number analyzed (Participants) | 440 | 211
  Week 24 | 64.1 | 69.2
  Week 36: number analyzed (Participants) | 430 | 204
  Week 36 | 67.2 | 71.6
  Week 48: number analyzed (Participants) | 422 | 199
  Week 48 | 65.9 | 65.3
  Week 60: number analyzed (Participants) | 398 | 187
  Week 60 | 67.3 | 66.3
  Week 72: number analyzed (Participants) | 387 | 173
  Week 72 | 68.5 | 65.9
  Week 84: number analyzed (Participants) | 376 | 170
  Week 84 | 69.9 | 73.5
  Week 96: number analyzed (Participants) | 377 | 164
  Week 96 | 73.2 | 69.5
  Week 108: number analyzed (Participants) | 357 | 159
  Week 108 | 68.3 | 66.7
  Week 120: number analyzed (Participants) | 332 | 157
  Week 120 | 72.9 | 67.5
  Week 132: number analyzed (Participants) | 331 | 153
  Week 132 | 71.3 | 66.7
  Week 144: number analyzed (Participants) | 327 | 154
  Week 144 | 71.3 | 67.5
  Week 156: number analyzed (Participants) | 290 | 135
  Week 156 | 72.4 | 63.0
  Week 168: number analyzed (Participants) | 297 | 138
  Week 168 | 73.4 | 60.9
  Week 180: number analyzed (Participants) | 292 | 140
  Week 180 | 72.6 | 67.1
  Week 192: number analyzed (Participants) | 283 | 134
  Week 192 | 67.5 | 67.9
  Week 204: number analyzed (Participants) | 270 | 134
  Week 204 | 69.6 | 69.4
  Week 216: number analyzed (Participants) | 263 | 132
  Week 216 | 68.1 | 64.4
  Week 228: number analyzed (Participants) | 265 | 126
  Week 228 | 72.1 | 66.7
  Week 240: number analyzed (Participants) | 254 | 118
  Week 240 | 66.9 | 69.5
  Week 252: number analyzed (Participants) | 232 | 111
  Week 252 | 68.5 | 71.2
  Week 264: number analyzed (Participants) | 228 | 107
  Week 264 | 66.7 | 74.8
  Week 276: number analyzed (Participants) | 216 | 114
  Week 276 | 68.1 | 76.3
  Week 288: number analyzed (Participants) | 209 | 110
  Week 288 | 70.8 | 73.6
  Week 300: number analyzed (Participants) | 200 | 105
  Week 300 | 72.5 | 66.7
  Week 312: number analyzed (Participants) | 207 | 101
  Week 312 | 69.6 | 64.4
  Week 324: number analyzed (Participants) | 205 | 104
  Week 324 | 72.7 | 65.4
  Week 336: number analyzed (Participants) | 194 | 97
  Week 336 | 70.1 | 63.9
  Week 348: number analyzed (Participants) | 188 | 92
  Week 348 | 71.8 | 69.6
  Week 360: number analyzed (Participants) | 180 | 86
  Week 360 | 67.8 | 67.4
  Week 372: number analyzed (Participants) | 167 | 83
  Week 372 | 70.7 | 71.1
  Week 384: number analyzed (Participants) | 165 | 80
  Week 384 | 64.2 | 65.0
  Week 396: number analyzed (Participants) | 151 | 77
  Week 396 | 65.6 | 64.9
  Week 408: number analyzed (Participants) | 3 | 2
  Week 408 | 66.7 | 50.0

6. Secondary Outcome: Percentage of Participants Achieving ACR70 Response: NRI
Description: The ACR response was a measurement of improvement in multiple disease assessment criteria.
  ACR70 response was defined as : 1) ≥ 70% improvement from baseline in SJC66, and 2) ≥ 70% improvement from baseline in TJC68, and 3) ≥ 70% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2.SGA (VAS), 3. PGA (VAS), 4. Total HAQ-DI score, and 5. hsCRP.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline | 30.0 | 23.1
  Week 12 | 36.8 | 36.4
  Week 24 | 37.8 | 39.3
  Week 36 | 40.6 | 37.2
  Week 48 | 39.4 | 36.4
  Week 60 | 36.4 | 34.3
  Week 72 | 38.0 | 30.2
  Week 84 | 36.8 | 34.3
  Week 96 | 39.6 | 28.1
  Week 108 | 35.4 | 29.8
  Week 120 | 36.0 | 31.0
  Week 132 | 32.8 | 29.3
  Week 144 | 31.6 | 28.5
  Week 156 | 26.8 | 22.3
  Week 168 | 30.8 | 24.0
  Week 180 | 30.8 | 25.6
  Week 192 | 26.6 | 25.2
  Week 204 | 26.6 | 24.8
  Week 216 | 26.4 | 23.1
  Week 228 | 27.2 | 24.4
  Week 240 | 21.5 | 21.5
  Week 252 | 21.7 | 20.7
  Week 264 | 23.1 | 22.7
  Week 276 | 21.3 | 24.8
  Week 288 | 22.1 | 24.8
  Week 300 | 22.5 | 19.8
  Week 312 | 23.1 | 19.8
  Week 324 | 21.5 | 21.1
  Week 336 | 20.3 | 17.8
  Week 348 | 19.7 | 19.0
  Week 360 | 17.7 | 16.1
  Week 372 | 16.7 | 17.4
  Week 384 | 14.9 | 14.9
  Week 396 | 14.9 | 14.5
  Week 408 | 0.4 | 0.4

7. Secondary Outcome: Percentage of Participants Achieving ACR70 Response: OC
Description: The ACR response was a measurement of improvement in multiple disease assessment criteria.
  ACR70 response was defined as : 1) ≥ 70% improvement from baseline in SJC66, and 2) ≥ 70% improvement from baseline in TJC68, and 3) ≥ 70% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2.SGA (VAS), 3. PGA (VAS), 4. Total HAQ-DI score, and 5.hsCRP.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline: number analyzed (Participants) | 491 | 238
  Extension Baseline | 30.3 | 23.5
  Week 12: number analyzed (Participants) | 486 | 231
  Week 12 | 37.7 | 38.1
  Week 24: number analyzed (Participants) | 440 | 211
  Week 24 | 42.7 | 45.0
  Week 36: number analyzed (Participants) | 431 | 202
  Week 36 | 46.9 | 44.6
  Week 48: number analyzed (Participants) | 421 | 200
  Week 48 | 46.6 | 44.0
  Week 60: number analyzed (Participants) | 398 | 186
  Week 60 | 45.5 | 44.6
  Week 72: number analyzed (Participants) | 388 | 173
  Week 72 | 48.7 | 42.2
  Week 84: number analyzed (Participants) | 374 | 171
  Week 84 | 48.9 | 48.5
  Week 96: number analyzed (Participants) | 375 | 165
  Week 96 | 52.5 | 41.2
  Week 108: number analyzed (Participants) | 354 | 159
  Week 108 | 49.7 | 45.3
  Week 120: number analyzed (Participants) | 333 | 158
  Week 120 | 53.8 | 47.5
  Week 132: number analyzed (Participants) | 333 | 153
  Week 132 | 48.9 | 46.4
  Week 144: number analyzed (Participants) | 325 | 156
  Week 144 | 48.3 | 44.2
  Week 156: number analyzed (Participants) | 292 | 135
  Week 156 | 45.5 | 40.0
  Week 168: number analyzed (Participants) | 297 | 136
  Week 168 | 51.5 | 42.6
  Week 180: number analyzed (Participants) | 292 | 141
  Week 180 | 52.4 | 44.0
  Week 192: number analyzed (Participants) | 283 | 135
  Week 192 | 46.6 | 45.2
  Week 204: number analyzed (Participants) | 269 | 133
  Week 204 | 49.1 | 45.1
  Week 216: number analyzed (Participants) | 265 | 132
  Week 216 | 49.4 | 42.4
  Week 228: number analyzed (Participants) | 265 | 126
  Week 228 | 50.9 | 46.8
  Week 240: number analyzed (Participants) | 254 | 120
  Week 240 | 42.1 | 43.3
  Week 252: number analyzed (Participants) | 233 | 110
  Week 252 | 46.4 | 45.5
  Week 264: number analyzed (Participants) | 227 | 107
  Week 264 | 50.7 | 51.4
  Week 276: number analyzed (Participants) | 217 | 113
  Week 276 | 48.8 | 53.1
  Week 288: number analyzed (Participants) | 210 | 110
  Week 288 | 52.4 | 54.5
  Week 300: number analyzed (Participants) | 202 | 105
  Week 300 | 55.4 | 45.7
  Week 312: number analyzed (Participants) | 208 | 101
  Week 312 | 55.3 | 47.5
  Week 324: number analyzed (Participants) | 205 | 104
  Week 324 | 52.2 | 49.0
  Week 336: number analyzed (Participants) | 195 | 97
  Week 336 | 51.8 | 44.3
  Week 348: number analyzed (Participants) | 190 | 92
  Week 348 | 51.6 | 50.0
  Week 360: number analyzed (Participants) | 179 | 87
  Week 360 | 49.2 | 44.8
  Week 372: number analyzed (Participants) | 169 | 84
  Week 372 | 49.1 | 50.0
  Week 384: number analyzed (Participants) | 163 | 80
  Week 384 | 45.4 | 45.0
  Week 396: number analyzed (Participants) | 151 | 77
  Week 396 | 49.0 | 45.5
  Week 408: number analyzed (Participants) | 3 | 2
  Week 408 | 66.7 | 50.0

8. Secondary Outcome: ACR N% Improvement (ACR-N) Response: OC
Description: ACR-N was defined as the smallest percentage improvement from core baseline in SJC66, TJC68 and the median of the following 5 items (Pain VAS [taken from the HAQ-DI], 2.SGA (VAS), 3. PGA (VAS), 4. Total HAQ-DI score, and 5. hsCRP). It had a range between 0 and 100%.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of improvement
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of improvement
  Extension Baseline: number analyzed (Participants) | 482 | 227
  Extension Baseline | 48.1 (30.29) | 46.3 (27.77)
  Week 12: number analyzed (Participants) | 478 | 226
  Week 12 | 56.3 (28.43) | 56.3 (27.13)
  Week 24: number analyzed (Participants) | 435 | 205
  Week 24 | 57.9 (29.64) | 60.8 (27.76)
  Week 36: number analyzed (Participants) | 424 | 201
  Week 36 | 59.8 (29.70) | 60.7 (27.95)
  Week 48: number analyzed (Participants) | 413 | 196
  Week 48 | 59.6 (30.69) | 58.9 (28.65)
  Week 60: number analyzed (Participants) | 388 | 181
  Week 60 | 59.9 (29.97) | 60.1 (28.43)
  Week 72: number analyzed (Participants) | 379 | 169
  Week 72 | 61.4 (28.92) | 59.0 (28.47)
  Week 84: number analyzed (Participants) | 367 | 168
  Week 84 | 61.6 (29.07) | 63.6 (26.74)
  Week 96: number analyzed (Participants) | 370 | 161
  Week 96 | 64.8 (28.61) | 61.2 (26.87)
  Week 108: number analyzed (Participants) | 348 | 156
  Week 108 | 61.2 (30.22) | 60.9 (28.69)
  Week 120: number analyzed (Participants) | 327 | 155
  Week 120 | 63.4 (29.25) | 61.1 (28.72)
  Week 132: number analyzed (Participants) | 325 | 147
  Week 132 | 62.3 (29.15) | 61.3 (28.52)
  Week 144: number analyzed (Participants) | 317 | 152
  Week 144 | 61.7 (28.99) | 60.8 (29.12)
  Week 156: number analyzed (Participants) | 280 | 132
  Week 156 | 61.5 (28.05) | 58.0 (27.70)
  Week 168: number analyzed (Participants) | 283 | 135
  Week 168 | 62.8 (29.75) | 56.9 (30.25)
  Week 180: number analyzed (Participants) | 283 | 138
  Week 180 | 63.2 (28.29) | 59.9 (29.79)
  Week 192: number analyzed (Participants) | 276 | 131
  Week 192 | 60.4 (29.15) | 61.5 (27.30)
  Week 204: number analyzed (Participants) | 264 | 131
  Week 204 | 62.3 (28.64) | 61.9 (26.79)
  Week 216: number analyzed (Participants) | 256 | 130
  Week 216 | 61.6 (29.87) | 61.4 (26.86)
  Week 228: number analyzed (Participants) | 259 | 124
  Week 228 | 64.2 (27.83) | 63.0 (26.45)
  Week 240: number analyzed (Participants) | 251 | 117
  Week 240 | 59.8 (28.22) | 60.6 (28.48)
  Week 252: number analyzed (Participants) | 227 | 107
  Week 252 | 62.4 (28.71) | 62.5 (26.24)
  Week 264: number analyzed (Participants) | 221 | 106
  Week 264 | 63.4 (29.81) | 64.4 (27.05)
  Week 276: number analyzed (Participants) | 209 | 111
  Week 276 | 63.3 (28.27) | 65.9 (25.42)
  Week 288: number analyzed (Participants) | 203 | 107
  Week 288 | 65.1 (29.68) | 63.0 (29.82)
  Week 300: number analyzed (Participants) | 196 | 103
  Week 300 | 64.9 (30.16) | 61.9 (27.14)
  Week 312: number analyzed (Participants) | 202 | 99
  Week 312 | 64.8 (29.89) | 59.9 (30.37)
  Week 324: number analyzed (Participants) | 197 | 101
  Week 324 | 65.9 (27.39) | 61.2 (30.98)
  Week 336: number analyzed (Participants) | 189 | 94
  Week 336 | 62.7 (29.35) | 59.8 (28.90)
  Week 348: number analyzed (Participants) | 181 | 91
  Week 348 | 64.8 (29.26) | 62.8 (28.29)
  Week 360: number analyzed (Participants) | 170 | 80
  Week 360 | 62.7 (29.81) | 61.2 (28.32)
  Week 372: number analyzed (Participants) | 152 | 70
  Week 372 | 64.2 (28.58) | 64.6 (29.43)
  Week 384: number analyzed (Participants) | 151 | 63
  Week 384 | 60.0 (30.27) | 62.9 (30.43)
  Week 396: number analyzed (Participants) | 135 | 57
  Week 396 | 61.5 (31.34) | 64.7 (28.98)
  Week 408: number analyzed (Participants) | 3 | 2
  Week 408 | 65.9 (41.08) | 35.4 (50.04)

9. Secondary Outcome: Change From Core Baseline in Disease Activity Score Based on 28 Joints Using C-reactive Protein (DAS28[CRP]): OC
Description: The DAS28(CRP) was a measure of the participant's disease activity calculated using the TJC (28 joints), SJC (28 joints), SGA [using a VAS on a scale of 0 (very well) to 100 (very poor)] and hsCRP using the formula:
  DAS28(CRP) = 0.56 * Square root [SQRT] (TJC28) + 0.28 * SQRT(SJC28) + 0.36 * Ln(CRP+1) + 0.014 * SGA + 0.96
  and the total possible score ranged from 1 to 9.4. Higher values indicated higher disease activity. A negative change from baseline indicated improvement.
Time Frame: Core Baseline, Extension Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, 384, 396, 408
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 491 | 234
  Change from Core Baseline at Extension Baseline | -2.7 (1.40) | -2.6 (1.28)
  Change from Core Baseline at Week 12: number analyzed (Participants) | 487 | 232
  Change from Core Baseline at Week 12 | -3.1 (1.28) | -3.1 (1.22)
  Change from Core Baseline at Week 24: number analyzed (Participants) | 443 | 211
  Change from Core Baseline at Week 24 | -3.2 (1.29) | -3.2 (1.33)
  Change from Core Baseline at Week 36: number analyzed (Participants) | 434 | 206
  Change from Core Baseline at Week 36 | -3.3 (1.28) | -3.3 (1.22)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 421 | 201
  Change from Core Baseline at Week 48 | -3.3 (1.32) | -3.3 (1.26)
  Change from Core Baseline at Week 60: number analyzed (Participants) | 398 | 187
  Change from Core Baseline at Week 60 | -3.3 (1.22) | -3.4 (1.17)
  Change from Core Baseline at Week 72: number analyzed (Participants) | 386 | 173
  Change from Core Baseline at Week 72 | -3.3 (1.23) | -3.4 (1.21)
  Change from Core Baseline at Week 84: number analyzed (Participants) | 377 | 172
  Change from Core Baseline at Week 84 | -3.4 (1.21) | -3.5 (1.09)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 377 | 165
  Change from Core Baseline at Week 96 | -3.4 (1.22) | -3.4 (1.13)
  Change from Core Baseline at Week 108: number analyzed (Participants) | 356 | 159
  Change from Core Baseline at Week 108 | -3.4 (1.22) | -3.3 (1.21)
  Change from Core Baseline at Week 120: number analyzed (Participants) | 334 | 159
  Change from Core Baseline at Week 120 | -3.4 (1.20) | -3.5 (1.14)
  Change from Core Baseline at Week 132: number analyzed (Participants) | 333 | 153
  Change from Core Baseline at Week 132 | -3.3 (1.21) | -3.5 (1.26)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 325 | 157
  Change from Core Baseline at Week 144 | -3.4 (1.19) | -3.4 (1.15)
  Change from Core Baseline at Week 156: number analyzed (Participants) | 290 | 136
  Change from Core Baseline at Week 156 | -3.4 (1.22) | -3.4 (1.28)
  Change from Core Baseline at Week 168: number analyzed (Participants) | 297 | 139
  Change from Core Baseline at Week 168 | -3.4 (1.27) | -3.4 (1.20)
  Change from Core Baseline at Week 180: number analyzed (Participants) | 292 | 143
  Change from Core Baseline at Week 180 | -3.4 (1.12) | -3.4 (1.21)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 285 | 135
  Change from Core Baseline at Week 192 | -3.3 (1.16) | -3.5 (1.13)
  Change from Core Baseline at Week 204: number analyzed (Participants) | 273 | 135
  Change from Core Baseline at Week 204 | -3.4 (1.16) | -3.5 (1.06)
  Change from Core Baseline at Week 216: number analyzed (Participants) | 264 | 133
  Change from Core Baseline at Week 216 | -3.4 (1.16) | -3.5 (1.15)
  Change from Core Baseline at Week 228: number analyzed (Participants) | 267 | 127
  Change from Core Baseline at Week 228 | -3.5 (1.12) | -3.5 (1.09)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 257 | 122
  Change from Core Baseline at Week 240 | -3.4 (1.13) | -3.4 (1.19)
  Change from Core Baseline at Week 252: number analyzed (Participants) | 233 | 109
  Change from Core Baseline at Week 252 | -3.5 (1.11) | -3.6 (1.24)
  Change from Core Baseline at Week 264: number analyzed (Participants) | 227 | 110
  Change from Core Baseline at Week 264 | -3.5 (1.19) | -3.6 (1.20)
  Change from Core Baseline at Week 276: number analyzed (Participants) | 215 | 114
  Change from Core Baseline at Week 276 | -3.5 (1.10) | -3.6 (1.17)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 208 | 111
  Change from Core Baseline at Week 288 | -3.5 (1.22) | -3.6 (1.28)
  Change from Core Baseline at Week 300: number analyzed (Participants) | 202 | 106
  Change from Core Baseline at Week 300 | -3.6 (1.19) | -3.5 (1.23)
  Change from Core Baseline at Week 312: number analyzed (Participants) | 207 | 101
  Change from Core Baseline at Week 312 | -3.5 (1.27) | -3.4 (1.30)
  Change from Core Baseline at Week 324: number analyzed (Participants) | 202 | 103
  Change from Core Baseline at Week 324 | -3.6 (1.14) | -3.5 (1.24)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 194 | 96
  Change from Core Baseline at Week 336 | -3.5 (1.17) | -3.4 (1.16)
  Change from Core Baseline at Week 348: number analyzed (Participants) | 186 | 93
  Change from Core Baseline at Week 348 | -3.5 (1.20) | -3.6 (1.14)
  Change from Core Baseline at Week 360: number analyzed (Participants) | 176 | 82
  Change from Core Baseline at Week 360 | -3.6 (1.21) | -3.4 (1.13)
  Change from Core Baseline at Week 372: number analyzed (Participants) | 155 | 72
  Change from Core Baseline at Week 372 | -3.6 (1.18) | -3.6 (1.26)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 155 | 64
  Change from Core Baseline at Week 384 | -3.4 (1.24) | -3.5 (1.26)
  Change from Core Baseline at Week 396: number analyzed (Participants) | 138 | 58
  Change from Core Baseline at Week 396 | -3.5 (1.38) | -3.8 (1.12)
  Change from Core Baseline at Week 408: number analyzed (Participants) | 3 | 2
  Change from Core Baseline at Week 408 | -3.8 (0.97) | -2.8 (0.25)

10. Secondary Outcome: Change From Core Baseline in Simple Disease Activity Index (SDAI): OC
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA (0 to 10 cm), PGA (0 to 10 cm), CRP (mg/dL). SDAI = TJC + SJC + SGA + PGA+ CRP. The SDAI score ranged from 0 to approximately 86. Higher SDAI indicated greater disease activity. A negative change from baseline indicated improvement.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 490 | 230
  Change from Core Baseline at Extension Baseline | -30.2 (15.49) | -29.8 (14.27)
  Change from Core Baseline at Week 12: number analyzed (Participants) | 485 | 228
  Change from Core Baseline at Week 12 | -33.4 (14.16) | -34.1 (13.79)
  Change from Core Baseline at Week 24: number analyzed (Participants) | 442 | 207
  Change from Core Baseline at Week 24 | -34.0 (14.19) | -35.0 (14.65)
  Change from Core Baseline at Week 36: number analyzed (Participants) | 432 | 203
  Change from Core Baseline at Week 36 | -34.7 (13.98) | -35.9 (13.42)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 420 | 197
  Change from Core Baseline at Week 48 | -34.7 (14.38) | -36.2 (14.08)
  Change from Core Baseline at Week 60: number analyzed (Participants) | 397 | 182
  Change from Core Baseline at Week 60 | -35.3 (13.57) | -36.3 (12.85)
  Change from Core Baseline at Week 72: number analyzed (Participants) | 385 | 170
  Change from Core Baseline at Week 72 | -35.4 (13.38) | -36.7 (13.41)
  Change from Core Baseline at Week 84: number analyzed (Participants) | 374 | 169
  Change from Core Baseline at Week 84 | -35.6 (13.38) | -37.3 (13.12)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 376 | 162
  Change from Core Baseline at Week 96 | -36.2 (13.31) | -36.8 (13.47)
  Change from Core Baseline at Week 108: number analyzed (Participants) | 354 | 157
  Change from Core Baseline at Week 108 | -36.0 (13.56) | -36.6 (13.65)
  Change from Core Baseline at Week 120: number analyzed (Participants) | 332 | 156
  Change from Core Baseline at Week 120 | -36.1 (13.28) | -37.4 (12.90)
  Change from Core Baseline at Week 132: number analyzed (Participants) | 332 | 148
  Change from Core Baseline at Week 132 | -35.6 (13.38) | -36.9 (14.25)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 323 | 154
  Change from Core Baseline at Week 144 | -35.7 (13.15) | -36.9 (13.12)
  Change from Core Baseline at Week 156: number analyzed (Participants) | 288 | 134
  Change from Core Baseline at Week 156 | -35.5 (13.36) | -36.9 (14.46)
  Change from Core Baseline at Week 168: number analyzed (Participants) | 295 | 136
  Change from Core Baseline at Week 168 | -35.8 (14.18) | -36.9 (13.84)
  Change from Core Baseline at Week 180: number analyzed (Participants) | 291 | 140
  Change from Core Baseline at Week 180 | -36.2 (12.72) | -36.9 (13.33)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 283 | 132
  Change from Core Baseline at Week 192 | -35.5 (12.74) | -38.2 (13.66)
  Change from Core Baseline at Week 204: number analyzed (Participants) | 272 | 133
  Change from Core Baseline at Week 204 | -35.8 (12.78) | -38.5 (13.72)
  Change from Core Baseline at Week 216: number analyzed (Participants) | 262 | 131
  Change from Core Baseline at Week 216 | -36.1 (12.92) | -38.0 (13.85)
  Change from Core Baseline at Week 228: number analyzed (Participants) | 265 | 125
  Change from Core Baseline at Week 228 | -36.8 (12.38) | -37.9 (12.87)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 256 | 119
  Change from Core Baseline at Week 240 | -35.9 (12.69) | -37.1 (14.38)
  Change from Core Baseline at Week 252: number analyzed (Participants) | 232 | 108
  Change from Core Baseline at Week 252 | -37.2 (12.63) | -38.6 (14.85)
  Change from Core Baseline at Week 264: number analyzed (Participants) | 226 | 107
  Change from Core Baseline at Week 264 | -37.3 (12.98) | -39.2 (14.59)
  Change from Core Baseline at Week 276: number analyzed (Participants) | 214 | 112
  Change from Core Baseline at Week 276 | -37.5 (12.18) | -38.6 (13.98)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 207 | 108
  Change from Core Baseline at Week 288 | -37.0 (13.22) | -38.6 (15.09)
  Change from Core Baseline at Week 300: number analyzed (Participants) | 201 | 103
  Change from Core Baseline at Week 300 | -37.5 (13.55) | -38.0 (15.38)
  Change from Core Baseline at Week 312: number analyzed (Participants) | 206 | 99
  Change from Core Baseline at Week 312 | -37.1 (13.71) | -37.7 (15.54)
  Change from Core Baseline at Week 324: number analyzed (Participants) | 201 | 101
  Change from Core Baseline at Week 324 | -37.7 (13.06) | -38.1 (15.56)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 193 | 94
  Change from Core Baseline at Week 336 | -36.7 (12.52) | -36.6 (14.36)
  Change from Core Baseline at Week 348: number analyzed (Participants) | 185 | 91
  Change from Core Baseline at Week 348 | -37.0 (12.53) | -37.2 (13.02)
  Change from Core Baseline at Week 360: number analyzed (Participants) | 175 | 80
  Change from Core Baseline at Week 360 | -37.4 (12.83) | -36.3 (13.05)
  Change from Core Baseline at Week 372: number analyzed (Participants) | 155 | 70
  Change from Core Baseline at Week 372 | -37.3 (12.68) | -37.8 (13.64)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 155 | 63
  Change from Core Baseline at Week 384 | -36.5 (12.64) | -36.5 (14.58)
  Change from Core Baseline at Week 396: number analyzed (Participants) | 138 | 57
  Change from Core Baseline at Week 396 | -36.3 (14.32) | -39.5 (13.50)
  Change from Core Baseline at Week 408: number analyzed (Participants) | 3 | 2
  Change from Core Baseline at Week 408 | -40.4 (12.91) | -35.6 (5.98)

11. Secondary Outcome: Change From Core Baseline in Clinical Disease Activity Index (CDAI): OC
Description: The CDAI was the SDAI modified that excluded CRP and consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA (0 to 10 cm), PGA (0 to 10 cm). SDAI = TJC + SJC + SGA+ PGA. The CDAI score ranged from 0 to approximately 76. Higher CDAI indicated greater disease activity. A negative change from baseline indicated improvement.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 490 | 233
  Change from Core Baseline at Extension Baseline | -28.8 (14.58) | -28.0 (13.68)
  Change from Core Baseline at Week 12: number analyzed (Participants) | 486 | 229
  Change from Core Baseline at Week 12 | -31.8 (13.45) | -32.4 (12.76)
  Change from Core Baseline at Week 24: number analyzed (Participants) | 442 | 207
  Change from Core Baseline at Week 24 | -32.4 (13.63) | -32.9 (13.79)
  Change from Core Baseline at Week 36: number analyzed (Participants) | 432 | 203
  Change from Core Baseline at Week 36 | -33.0 (13.44) | -33.8 (12.51)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 421 | 197
  Change from Core Baseline at Week 48 | -33.1 (13.79) | -34.1 (13.18)
  Change from Core Baseline at Week 60: number analyzed (Participants) | 399 | 183
  Change from Core Baseline at Week 60 | -33.7 (12.97) | -34.2 (12.22)
  Change from Core Baseline at Week 72: number analyzed (Participants) | 386 | 170
  Change from Core Baseline at Week 72 | -33.8 (12.73) | -34.4 (12.57)
  Change from Core Baseline at Week 84: number analyzed (Participants) | 374 | 169
  Change from Core Baseline at Week 84 | -33.9 (12.82) | -35.2 (12.31)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 377 | 162
  Change from Core Baseline at Week 96 | -34.6 (12.76) | -34.7 (12.56)
  Change from Core Baseline at Week 108: number analyzed (Participants) | 355 | 157
  Change from Core Baseline at Week 108 | -34.3 (12.96) | -34.5 (12.92)
  Change from Core Baseline at Week 120: number analyzed (Participants) | 332 | 156
  Change from Core Baseline at Week 120 | -34.5 (12.70) | -35.2 (11.87)
  Change from Core Baseline at Week 132: number analyzed (Participants) | 333 | 148
  Change from Core Baseline at Week 132 | -34.1 (12.82) | -34.7 (13.07)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 323 | 154
  Change from Core Baseline at Week 144 | -34.1 (12.63) | -34.9 (12.12)
  Change from Core Baseline at Week 156: number analyzed (Participants) | 290 | 134
  Change from Core Baseline at Week 156 | -34.0 (12.74) | -34.8 (13.29)
  Change from Core Baseline at Week 168: number analyzed (Participants) | 297 | 136
  Change from Core Baseline at Week 168 | -34.1 (13.64) | -34.8 (12.55)
  Change from Core Baseline at Week 180: number analyzed (Participants) | 291 | 140
  Change from Core Baseline at Week 180 | -34.5 (12.10) | -34.8 (12.39)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 283 | 132
  Change from Core Baseline at Week 192 | -33.9 (12.10) | -35.9 (12.65)
  Change from Core Baseline at Week 204: number analyzed (Participants) | 272 | 133
  Change from Core Baseline at Week 204 | -34.2 (12.26) | -36.3 (12.79)
  Change from Core Baseline at Week 216: number analyzed (Participants) | 262 | 131
  Change from Core Baseline at Week 216 | -34.5 (12.18) | -36.0 (13.00)
  Change from Core Baseline at Week 228: number analyzed (Participants) | 265 | 125
  Change from Core Baseline at Week 228 | -35.2 (11.69) | -35.8 (11.98)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 256 | 119
  Change from Core Baseline at Week 240 | -34.3 (11.99) | -35.2 (13.27)
  Change from Core Baseline at Week 252: number analyzed (Participants) | 235 | 109
  Change from Core Baseline at Week 252 | -35.3 (11.94) | -36.4 (13.55)
  Change from Core Baseline at Week 264: number analyzed (Participants) | 227 | 108
  Change from Core Baseline at Week 264 | -35.6 (12.15) | -36.9 (13.53)
  Change from Core Baseline at Week 276: number analyzed (Participants) | 216 | 113
  Change from Core Baseline at Week 276 | -35.9 (11.38) | -36.4 (12.84)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 208 | 108
  Change from Core Baseline at Week 288 | -35.4 (12.28) | -36.5 (13.47)
  Change from Core Baseline at Week 300: number analyzed (Participants) | 201 | 103
  Change from Core Baseline at Week 300 | -35.8 (12.84) | -35.7 (14.29)
  Change from Core Baseline at Week 312: number analyzed (Participants) | 207 | 99
  Change from Core Baseline at Week 312 | -35.5 (13.10) | -35.5 (14.40)
  Change from Core Baseline at Week 324: number analyzed (Participants) | 202 | 102
  Change from Core Baseline at Week 324 | -35.8 (12.30) | -36.0 (14.37)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 195 | 96
  Change from Core Baseline at Week 336 | -35.0 (11.76) | -34.2 (13.32)
  Change from Core Baseline at Week 348: number analyzed (Participants) | 187 | 91
  Change from Core Baseline at Week 348 | -35.3 (11.70) | -34.8 (11.73)
  Change from Core Baseline at Week 360: number analyzed (Participants) | 180 | 86
  Change from Core Baseline at Week 360 | -35.5 (12.00) | -34.0 (11.54)
  Change from Core Baseline at Week 372: number analyzed (Participants) | 168 | 83
  Change from Core Baseline at Week 372 | -35.4 (12.46) | -33.9 (12.73)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 166 | 83
  Change from Core Baseline at Week 384 | -34.8 (11.82) | -32.6 (13.11)
  Change from Core Baseline at Week 396: number analyzed (Participants) | 154 | 79
  Change from Core Baseline at Week 396 | -34.7 (13.28) | -34.2 (12.55)
  Change from Core Baseline at Week 408: number analyzed (Participants) | 3 | 2
  Change from Core Baseline at Week 408 | -39.2 (12.87) | -34.9 (6.36)

12. Secondary Outcome: Percentage of Participants Achieving European League Against Rheumatism (EULAR) Response: OC
Description: DAS28(CRP) was categorized into EULAR response categories (none, moderate, good) as follows:
  None= Actual DAS28(CRP) ≤ 3.2, > 3.2 to ≤ 5.1, or > 5.1 AND Improvement in DAS28(CRP) from baseline ≤ 6.0 or > 0.6 to ≤ 1.2;
  Moderate= Actual DAS28(CRP) ≤ 3.2 AND Improvement in DAS28(CRP) from baseline > 0.6 to ≤ 1.2, Actual DAS28(CRP) > 3.2 to ≤ 5.1 or > 5.1 AND Improvement in DAS28(CRP) from baseline > 1.2, or Actual DAS28(CRP) > 3.2 to ≤ 5.1 AND Improvement in DAS28(CRP) from baseline > 0.6 to ≤ 1.2;
  Good= Actual DAS28(CRP) ≤ 3.2 AND Improvement in DAS28(CRP) from baseline > 1.2.
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline: Good: number analyzed (Participants) | 491 | 234
  Extension Baseline: Good | 46.2 | 41.5
  Extension Baseline: Moderate: number analyzed (Participants) | 491 | 234
  Extension Baseline: Moderate | 43.6 | 48.7
  Extension Baseline: None: number analyzed (Participants) | 491 | 234
  Extension Baseline: None | 10.2 | 9.8
  Week 12: Good: number analyzed (Participants) | 487 | 232
  Week 12: Good | 59.1 | 60.3
  Week 12: Moderate: number analyzed (Participants) | 487 | 232
  Week 12: Moderate | 35.5 | 34.9
  Week 12: None: number analyzed (Participants) | 487 | 232
  Week 12: None | 5.3 | 4.7
  Week 24: Good: number analyzed (Participants) | 443 | 211
  Week 24: Good | 65.2 | 65.9
  Week 24: Moderate: number analyzed (Participants) | 443 | 211
  Week 24: Moderate | 29.3 | 28.9
  Week 24: None: number analyzed (Participants) | 443 | 211
  Week 24: None | 5.4 | 5.2
  Week 36: Good: number analyzed (Participants) | 434 | 206
  Week 36: Good | 66.4 | 66.0
  Week 36: Moderate: number analyzed (Participants) | 434 | 206
  Week 36: Moderate | 29.7 | 30.6
  Week 36: None: number analyzed (Participants) | 434 | 206
  Week 36: None | 3.9 | 3.4
  Week 48: Good: number analyzed (Participants) | 421 | 201
  Week 48: Good | 67.7 | 68.7
  Week 48: Moderate: number analyzed (Participants) | 421 | 201
  Week 48: Moderate | 27.8 | 27.4
  Week 48: None: number analyzed (Participants) | 421 | 201
  Week 48: None | 4.5 | 4.0
  Week 60: Good: number analyzed (Participants) | 398 | 187
  Week 60: Good | 67.8 | 64.2
  Week 60: Moderate: number analyzed (Participants) | 398 | 187
  Week 60: Moderate | 29.9 | 34.2
  Week 60: None: number analyzed (Participants) | 398 | 187
  Week 60: None | 2.3 | 1.6
  Week 72: Good: number analyzed (Participants) | 386 | 173
  Week 72: Good | 70.5 | 65.3
  Week 72: Moderate: number analyzed (Participants) | 386 | 173
  Week 72: Moderate | 26.7 | 32.9
  Week 72: None: number analyzed (Participants) | 386 | 173
  Week 72: None | 2.8 | 1.7
  Week 84: Good: number analyzed (Participants) | 377 | 172
  Week 84: Good | 70.3 | 69.8
  Week 84: Moderate: number analyzed (Participants) | 377 | 172
  Week 84: Moderate | 27.6 | 29.1
  Week 84: None: number analyzed (Participants) | 377 | 172
  Week 84: None | 2.1 | 1.2
  Week 96: Good: number analyzed (Participants) | 377 | 165
  Week 96: Good | 72.9 | 69.1
  Week 96: Moderate: number analyzed (Participants) | 377 | 165
  Week 96: Moderate | 25.2 | 27.9
  Week 96: None: number analyzed (Participants) | 377 | 165
  Week 96: None | 1.9 | 3.0
  Week 108: Good: number analyzed (Participants) | 356 | 159
  Week 108: Good | 74.2 | 66.7
  Week 108: Moderate: number analyzed (Participants) | 356 | 159
  Week 108: Moderate | 23.6 | 29.6
  Week 108: None: number analyzed (Participants) | 356 | 159
  Week 108: None | 2.2 | 3.8
  Week 120: Good: number analyzed (Participants) | 334 | 159
  Week 120: Good | 74.6 | 67.9
  Week 120: Moderate: number analyzed (Participants) | 334 | 159
  Week 120: Moderate | 23.7 | 29.6
  Week 120: None: number analyzed (Participants) | 334 | 159
  Week 120: None | 1.8 | 2.5
  Week 132: Good: number analyzed (Participants) | 333 | 153
  Week 132: Good | 69.1 | 69.9
  Week 132: Moderate: number analyzed (Participants) | 333 | 153
  Week 132: Moderate | 28.8 | 27.5
  Week 132: None: number analyzed (Participants) | 333 | 153
  Week 132: None | 2.1 | 2.6
  Week 144: Good: number analyzed (Participants) | 325 | 157
  Week 144: Good | 72.3 | 65.6
  Week 144: Moderate: number analyzed (Participants) | 325 | 157
  Week 144: Moderate | 25.8 | 33.1
  Week 144: None: number analyzed (Participants) | 325 | 157
  Week 144: None | 1.8 | 1.3
  Week 156: Good: number analyzed (Participants) | 290 | 136
  Week 156: Good | 69.0 | 64.7
  Week 156: Moderate: number analyzed (Participants) | 290 | 136
  Week 156: Moderate | 28.3 | 30.9
  Week 156: None: number analyzed (Participants) | 290 | 136
  Week 156: None | 2.8 | 4.4
  Week 168: Good: number analyzed (Participants) | 297 | 139
  Week 168: Good | 73.4 | 68.3
  Week 168: Moderate: number analyzed (Participants) | 297 | 139
  Week 168: Moderate | 23.6 | 29.5
  Week 168: None: number analyzed (Participants) | 297 | 139
  Week 168: None | 3.0 | 2.2
  Week 180: Good: number analyzed (Participants) | 292 | 143
  Week 180: Good | 74.0 | 68.5
  Week 180: Moderate: number analyzed (Participants) | 292 | 143
  Week 180: Moderate | 25.3 | 28.7
  Week 180: None: number analyzed (Participants) | 292 | 143
  Week 180: None | 0.7 | 2.8
  Week 192: Good: number analyzed (Participants) | 285 | 135
  Week 192: Good | 71.2 | 71.1
  Week 192: Moderate: number analyzed (Participants) | 285 | 135
  Week 192: Moderate | 26.3 | 28.1
  Week 192: None: number analyzed (Participants) | 285 | 135
  Week 192: None | 2.5 | 0.7
  Week 204: Good: number analyzed (Participants) | 273 | 135
  Week 204: Good | 73.3 | 76.3
  Week 204: Moderate: number analyzed (Participants) | 273 | 135
  Week 204: Moderate | 23.8 | 22.2
  Week 204: None: number analyzed (Participants) | 273 | 135
  Week 204: None | 2.9 | 1.5
  Week 216: Good: number analyzed (Participants) | 264 | 133
  Week 216: Good | 72.7 | 69.9
  Week 216: Moderate: number analyzed (Participants) | 264 | 133
  Week 216: Moderate | 26.1 | 28.6
  Week 216: None: number analyzed (Participants) | 264 | 133
  Week 216: None | 1.1 | 1.5
  Week 228: Good: number analyzed (Participants) | 267 | 127
  Week 228: Good | 76.4 | 70.1
  Week 228: Moderate: number analyzed (Participants) | 267 | 127
  Week 228: Moderate | 23.6 | 29.9
  Week 228: None: number analyzed (Participants) | 267 | 127
  Week 228: None | 0 | 0
  Week 240: Good: number analyzed (Participants) | 257 | 122
  Week 240: Good | 73.2 | 63.1
  Week 240: Moderate: number analyzed (Participants) | 257 | 122
  Week 240: Moderate | 26.1 | 36.9
  Week 240: None: number analyzed (Participants) | 257 | 122
  Week 240: None | 0.8 | 0
  Week 252: Good: number analyzed (Participants) | 233 | 109
  Week 252: Good | 74.2 | 73.4
  Week 252: Moderate: number analyzed (Participants) | 233 | 109
  Week 252: Moderate | 24.5 | 25.7
  Week 252: None: number analyzed (Participants) | 233 | 109
  Week 252: None | 1.3 | 0.9
  Week 264: Good: number analyzed (Participants) | 227 | 110
  Week 264: Good | 74.4 | 75.5
  Week 264: Moderate: number analyzed (Participants) | 227 | 110
  Week 264: Moderate | 24.2 | 22.7
  Week 264: None: number analyzed (Participants) | 227 | 110
  Week 264: None | 1.3 | 1.8
  Week 276: Good: number analyzed (Participants) | 215 | 114
  Week 276: Good | 74.4 | 70.2
  Week 276: Moderate: number analyzed (Participants) | 215 | 114
  Week 276: Moderate | 25.1 | 28.1
  Week 276: None: number analyzed (Participants) | 215 | 114
  Week 276: None | 0.5 | 1.8
  Week 288: Good: number analyzed (Participants) | 208 | 111
  Week 288: Good | 73.6 | 73.0
  Week 288: Moderate: number analyzed (Participants) | 208 | 111
  Week 288: Moderate | 24.5 | 24.3
  Week 288: None: number analyzed (Participants) | 208 | 111
  Week 288: None | 1.9 | 2.7
  Week 300: Good: number analyzed (Participants) | 202 | 106
  Week 300: Good | 74.8 | 74.5
  Week 300: Moderate: number analyzed (Participants) | 202 | 106
  Week 300: Moderate | 23.8 | 25.5
  Week 300: None: number analyzed (Participants) | 202 | 106
  Week 300: None | 1.5 | 0
  Week 312: Good: number analyzed (Participants) | 207 | 101
  Week 312: Good | 75.8 | 66.3
  Week 312: Moderate: number analyzed (Participants) | 207 | 101
  Week 312: Moderate | 22.2 | 32.7
  Week 312: None: number analyzed (Participants) | 207 | 101
  Week 312: None | 1.9 | 1.0
  Week 324: Good: number analyzed (Participants) | 202 | 103
  Week 324: Good | 75.7 | 71.8
  Week 324: Moderate: number analyzed (Participants) | 202 | 103
  Week 324: Moderate | 21.8 | 26.2
  Week 324: None: number analyzed (Participants) | 202 | 103
  Week 324: None | 2.5 | 1.9
  Week 336: Good: number analyzed (Participants) | 194 | 96
  Week 336: Good | 74.2 | 71.9
  Week 336: Moderate: number analyzed (Participants) | 194 | 96
  Week 336: Moderate | 24.7 | 26.0
  Week 336: None: number analyzed (Participants) | 194 | 96
  Week 336: None | 1.0 | 2.1
  Week 348: Good: number analyzed (Participants) | 186 | 93
  Week 348: Good | 76.9 | 78.5
  Week 348: Moderate: number analyzed (Participants) | 186 | 93
  Week 348: Moderate | 21.5 | 20.4
  Week 348: None: number analyzed (Participants) | 186 | 93
  Week 348: None | 1.6 | 1.1
  Week 360: Good: number analyzed (Participants) | 176 | 82
  Week 360: Good | 73.3 | 73.2
  Week 360: Moderate: number analyzed (Participants) | 176 | 82
  Week 360: Moderate | 23.9 | 24.4
  Week 360: None: number analyzed (Participants) | 176 | 82
  Week 360: None | 2.8 | 2.4
  Week 372: Good: number analyzed (Participants) | 155 | 72
  Week 372: Good | 76.8 | 77.8
  Week 372: Moderate: number analyzed (Participants) | 155 | 72
  Week 372: Moderate | 21.3 | 18.1
  Week 372: None: number analyzed (Participants) | 155 | 72
  Week 372: None | 1.9 | 4.2
  Week 384: Good: number analyzed (Participants) | 155 | 64
  Week 384: Good | 70.3 | 78.1
  Week 384: Moderate: number analyzed (Participants) | 155 | 64
  Week 384: Moderate | 28.4 | 20.3
  Week 384: None: number analyzed (Participants) | 155 | 64
  Week 384: None | 1.3 | 1.6
  Week 396: Good: number analyzed (Participants) | 138 | 58
  Week 396: Good | 73.2 | 81.0
  Week 396: Moderate: number analyzed (Participants) | 138 | 58
  Week 396: Moderate | 21.7 | 19.0
  Week 396: None: number analyzed (Participants) | 138 | 58
  Week 396: None | 5.1 | 0
  Week 408: Good: number analyzed (Participants) | 3 | 2
  Week 408: Good | 100.0 | 50.0
  Week 408: Moderate: number analyzed (Participants) | 3 | 2
  Week 408: Moderate | 0 | 50.0
  Week 408: None: number analyzed (Participants) | 3 | 2
  Week 408: None | 0 | 0

13. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission: NRI
Description: A participant's disease activity status was defined as being in remission when scores on the TJC28, SJC28, CRP (actual value in mg/dL) and SGA (cm) were all ≤ 1.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline | 10.1 | 7.4
  Week 12 | 13.1 | 11.6
  Week 24 | 14.9 | 15.3
  Week 36 | 15.3 | 14.5
  Week 48 | 17.7 | 14.0
  Week 60 | 15.5 | 12.4
  Week 72 | 15.5 | 12.0
  Week 84 | 15.1 | 12.4
  Week 96 | 18.3 | 11.2
  Week 108 | 14.9 | 10.7
  Week 120 | 12.3 | 13.2
  Week 132 | 12.1 | 12.8
  Week 144 | 10.5 | 9.9
  Week 156 | 10.9 | 8.3
  Week 168 | 13.9 | 7.9
  Week 180 | 10.3 | 11.2
  Week 192 | 10.1 | 10.7
  Week 204 | 11.1 | 9.5
  Week 216 | 11.5 | 7.9
  Week 228 | 11.9 | 9.9
  Week 240 | 8.9 | 7.4
  Week 252 | 7.8 | 7.9
  Week 264 | 11.3 | 7.4
  Week 276 | 8.9 | 9.5
  Week 288 | 10.1 | 9.9
  Week 300 | 10.9 | 8.7
  Week 312 | 10.5 | 7.9
  Week 324 | 9.5 | 10.3
  Week 336 | 8.5 | 7.4
  Week 348 | 9.1 | 9.1
  Week 360 | 9.3 | 6.2
  Week 372 | 8.2 | 6.6
  Week 384 | 6.6 | 4.5
  Week 396 | 7.8 | 5.4
  Week 408 | 0.4 | 0

14. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission: OC
Description: as for outcome 13
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
percentage of participants
  Extension Baseline: number analyzed (Participants) | 495 | 240
  Extension Baseline | 10.1 | 7.5
  Week 12: number analyzed (Participants) | 489 | 236
  Week 12 | 13.3 | 11.9
  Week 24: number analyzed (Participants) | 446 | 215
  Week 24 | 16.6 | 17.2
  Week 36: number analyzed (Participants) | 435 | 206
  Week 36 | 17.5 | 17.0
  Week 48: number analyzed (Participants) | 426 | 204
  Week 48 | 20.7 | 16.7
  Week 60: number analyzed (Participants) | 402 | 189
  Week 60 | 19.2 | 15.9
  Week 72: number analyzed (Participants) | 390 | 174
  Week 72 | 19.7 | 16.7
  Week 84: number analyzed (Participants) | 381 | 173
  Week 84 | 19.7 | 17.3
  Week 96: number analyzed (Participants) | 379 | 168
  Week 96 | 24.0 | 16.1
  Week 108: number analyzed (Participants) | 359 | 161
  Week 108 | 20.6 | 16.1
  Week 120: number analyzed (Participants) | 340 | 160
  Week 120 | 17.9 | 20.0
  Week 132: number analyzed (Participants) | 335 | 157
  Week 132 | 17.9 | 19.7
  Week 144: number analyzed (Participants) | 330 | 158
  Week 144 | 15.8 | 15.2
  Week 156: number analyzed (Participants) | 296 | 139
  Week 156 | 18.2 | 14.4
  Week 168: number analyzed (Participants) | 299 | 139
  Week 168 | 23.1 | 13.7
  Week 180: number analyzed (Participants) | 293 | 144
  Week 180 | 17.4 | 18.8
  Week 192: number analyzed (Participants) | 288 | 138
  Week 192 | 17.4 | 18.8
  Week 204: number analyzed (Participants) | 276 | 135
  Week 204 | 19.9 | 17.0
  Week 216: number analyzed (Participants) | 269 | 134
  Week 216 | 21.2 | 14.2
  Week 228: number analyzed (Participants) | 268 | 129
  Week 228 | 22.0 | 18.6
  Week 240: number analyzed (Participants) | 262 | 123
  Week 240 | 16.8 | 14.6
  Week 252: number analyzed (Participants) | 239 | 113
  Week 252 | 16.3 | 16.8
  Week 264: number analyzed (Participants) | 231 | 111
  Week 264 | 24.2 | 16.2
  Week 276: number analyzed (Participants) | 218 | 115
  Week 276 | 20.2 | 20.0
  Week 288: number analyzed (Participants) | 215 | 111
  Week 288 | 23.3 | 21.6
  Week 300: number analyzed (Participants) | 205 | 107
  Week 300 | 26.3 | 19.6
  Week 312: number analyzed (Participants) | 210 | 105
  Week 312 | 24.8 | 18.1
  Week 324: number analyzed (Participants) | 207 | 105
  Week 324 | 22.7 | 23.8
  Week 336: number analyzed (Participants) | 197 | 98
  Week 336 | 21.3 | 18.4
  Week 348: number analyzed (Participants) | 190 | 94
  Week 348 | 23.7 | 23.4
  Week 360: number analyzed (Participants) | 185 | 90
  Week 360 | 24.9 | 16.7
  Week 372: number analyzed (Participants) | 167 | 85
  Week 372 | 24.6 | 18.8
  Week 384: number analyzed (Participants) | 165 | 85
  Week 384 | 20.0 | 12.9
  Week 396: number analyzed (Participants) | 155 | 80
  Week 396 | 25.2 | 16.3
  Week 408: number analyzed (Participants) | 3 | 2
  Week 408 | 66.7 | 0

15. Secondary Outcome: Change From Core Baseline in Physical Component Score (PCS) of Quality of Life Using the Short Form-36 (SF-36) Scores: OC
Description: The health-related quality of life of the subject was assessed using the SF-36 with a 4-week recall period. This consists of 36 questions belonging to 8 domains in 2 components:
  * Physical well-being: 4 domains: physical functioning (10 items), role physical (4 items), bodily pain (2 items), and general health (GH) perceptions (5 items).
  * Mental well-being: 4 domains: vitality (4 items), social functioning (2 items), role emotional (3 items), and mental health (5 items).
  These scales were from 0 to 100 with higher scores indicating a better quality of life.
Time Frame: Core Baseline, Extension Baseline, Weeks 48, 96, 144, 192, 240, 288, 336, 384
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 490 | 237
  Change from Core Baseline at Extension Baseline | 9.2 (9.11) | 9.5 (8.85)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 480 | 227
  Change from Core Baseline at Week 48 | 11.3 (9.45) | 11.5 (8.74)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 377 | 168
  Change from Core Baseline at Week 96 | 12.2 (9.70) | 11.8 (8.87)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 332 | 153
  Change from Core Baseline at Week 144 | 11.8 (9.86) | 12.2 (9.21)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 289 | 140
  Change from Core Baseline at Week 192 | 11.2 (9.21) | 11.0 (9.40)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 263 | 125
  Change from Core Baseline at Week 240 | 10.9 (9.58) | 11.4 (9.29)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 215 | 109
  Change from Core Baseline at Week 288 | 13.0 (10.71) | 13.1 (9.50)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 204 | 104
  Change from Core Baseline at Week 336 | 12.8 (10.12) | 12.0 (8.79)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 175 | 90
  Change from Core Baseline at Week 384 | 11.5 (9.97) | 11.7 (8.00)

16. Secondary Outcome: Change From Core Baseline in MCS of Quality of Life Using the SF-36 Scores: OC
Description: as for outcome 15
Time Frame: Core Baseline, Extension Baseline, Weeks 48, 96, 144, 192, 240, 288, 336, 384
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 490 | 237
  Change from Core Baseline at Extension Baseline | 6.1 (9.67) | 7.1 (10.01)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 480 | 227
  Change from Core Baseline at Week 48 | 6.2 (10.52) | 6.8 (10.84)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 377 | 168
  Change from Core Baseline at Week 96 | 6.5 (10.54) | 6.7 (10.33)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 332 | 153
  Change from Core Baseline at Week 144 | 6.2 (10.72) | 6.6 (10.86)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 289 | 140
  Change from Core Baseline at Week 192 | 6.1 (11.47) | 7.5 (11.60)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 263 | 125
  Change from Core Baseline at Week 240 | 6.5 (11.11) | 7.7 (11.66)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 215 | 109
  Change from Core Baseline at Week 288 | 7.3 (11.49) | 8.2 (11.20)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 204 | 104
  Change from Core Baseline at Week 336 | 6.7 (10.49) | 6.6 (13.65)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 175 | 90
  Change from Core Baseline at Week 384 | 6.3 (11.23) | 8.0 (10.98)

17. Secondary Outcome: Change From Core Baseline in Quality of Life Using Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale: OC
Description: FACIT-Fatigue scale was a 13-item questionnaire, each scored on a 5-point scale: 0 (Not at all) to 4 (Very much). Negatively stated items were reversed by subtracting the response from "4" before being added to obtain a total score. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score), with a higher score indicating less fatigue. A positive change from baseline indicated better quality of life.
Time Frame: Core Baseline, Extension Baseline, Weeks 48, 96, 144, 192, 240, 288, 336, 384
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
Number analyzed (Participants) | 497 | 242
score on a scale
  Change from Core Baseline at Extension Baseline: number analyzed (Participants) | 490 | 237
  Change from Core Baseline at Extension Baseline | 10.7 (11.06) | 12.1 (10.71)
  Change from Core Baseline at Week 48: number analyzed (Participants) | 481 | 227
  Change from Core Baseline at Week 48 | 11.6 (11.16) | 12.7 (11.62)
  Change from Core Baseline at Week 96: number analyzed (Participants) | 377 | 168
  Change from Core Baseline at Week 96 | 12.0 (11.59) | 12.9 (10.97)
  Change from Core Baseline at Week 144: number analyzed (Participants) | 332 | 153
  Change from Core Baseline at Week 144 | 12.3 (11.31) | 13.2 (11.92)
  Change from Core Baseline at Week 192: number analyzed (Participants) | 289 | 140
  Change from Core Baseline at Week 192 | 11.7 (11.63) | 12.8 (11.96)
  Change from Core Baseline at Week 240: number analyzed (Participants) | 264 | 124
  Change from Core Baseline at Week 240 | 11.5 (11.52) | 12.5 (11.74)
  Change from Core Baseline at Week 288: number analyzed (Participants) | 215 | 109
  Change from Core Baseline at Week 288 | 13.4 (13.21) | 15.0 (12.03)
  Change from Core Baseline at Week 336: number analyzed (Participants) | 204 | 104
  Change from Core Baseline at Week 336 | 13.2 (12.18) | 13.8 (12.29)
  Change from Core Baseline at Week 384: number analyzed (Participants) | 175 | 90
  Change from Core Baseline at Week 384 | 12.6 (13.35) | 13.9 (10.76)

ADVERSE EVENTS:
Time Frame: From First dose to Week 437
Description: Safety Analysis Set. As per planned analysis, data was collected and analyzed based on the parent study i.e. DARWIN 1 and DARWIN 2. No comparison/collection/analysis was planned based on extension study dose as it was not considered meaningful.
Arm/Group | Filgotinib Darwin 1 | Filgotinib Darwin 2
All-Cause Mortality (participants affected / at risk) | 8/497 | 8/242
Serious Adverse Events (participants affected / at risk) | 84/497 | 48/242
Other Adverse Events (participants affected / at risk) | 386/497 | 189/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filgotinib Darwin 1 (N=497) | Filgotinib Darwin 2 (N=242)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Caplan's syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Electrocardiogram Q wave abnormal (Investigations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (9) | 3 (4)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filgotinib Darwin 1 (N=497) | Filgotinib Darwin 2 (N=242)
Blood cholesterol increased (Investigations) | 13 (18) | 23 (42)
Mycobacterium tuberculosis complex test positive (Investigations) | 58 (59) | 40 (40)
Lymphocyte count decreased (Investigations) | 20 (31) | 18 (38)
Blood creatinine increased (Investigations) | 13 (14) | 20 (25)
Hypertension (Vascular disorders) | 75 (83) | 27 (37)
Headache (Nervous system disorders) | 34 (45) | 26 (41)
Lymphopenia (Blood and lymphatic system disorders) | 45 (65) | 23 (33)
Diarrhoea (Gastrointestinal disorders) | 33 (40) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (41) | 10 (15)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 41 (78) | 15 (23)
Bronchitis (Infections and infestations) | 59 (86) | 19 (22)
COVID-19 (Infections and infestations) | 34 (37) | 10 (10)
Herpes zoster (Infections and infestations) | 29 (32) | 14 (14)
Gastroenteritis (Infections and infestations) | 29 (32) | 8 (10)
Influenza (Infections and infestations) | 30 (39) | 12 (16)
Nasopharyngitis (Infections and infestations) | 70 (112) | 24 (37)
Upper respiratory tract infection (Infections and infestations) | 57 (82) | 37 (50)
Pharyngitis (Infections and infestations) | 31 (41) | 11 (13)
Urinary tract infection (Infections and infestations) | 72 (128) | 30 (58)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 39 (54) | 30 (54)
Dyslipidaemia (Metabolism and nutrition disorders) | 39 (53) | 17 (22)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 18 (28) | 13 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02065700/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT02065700/SAP_001.pdf